CLINICAL TRIAL: NCT03456479
Title: Diagnosis of Cow's Milk Protein Allergy Among Infants and Children in Assuit University
Brief Title: Diagnosis of Cow's Milk Protein Allergy Among Infants and Children in Assuit University Children Hospital
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gamal Nady Rady Ibrahim, Assiut - Egypt, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: cow's milk protein allergy
Record Dates: First submitted 2018-03-03; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Cow Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: skin prick test - specific serum IgE — The study will assess the diagnosis of Cow's milk protein allergy (CMPA) among infant and children in Assiut University Children Hospital using skin prick test and specificserumIgE

SUMMARY:
The study will assess the diagnosis of Cow's milk protein allergy (CMPA) among infant and children in Assiut University Children Hospital using skin prick test and specific serum IgE

DETAILED DESCRIPTION:
Food allergy is a reproducible specific immune response to the exposure to a given food. Cow's milk protein allergy (CMPA) is a clinically abnormal reaction to cow's milk protein (CMP) via immune mechanisms triggered by milk protein (Boyce etal., 2010) .

According to the European Academy for Allergy and Clinical Immunology (EAACI) and the World Allergy Organization (WAO), a hypersensitivity reaction to cow's milk involving the immune system can be called as CMPA.There is difference between CMPA and non-allergic cow's milk intolerance (e.glactose intolerance) which occurs as a result of lactase deficiency without involvement of the immune system (Venter etal ., 2013) .

CMPA is categorized into immunoglobulin IgE mediated, non-IgE mediated, or mixed CMPA(Sichereretal ., 2001) .

1.9% to 4.9% prevalence of CMPA among children with a peak in prevalence (2-3%) in the first year of life and prevalence of <1% in children aged ≥6 years(Koletzkoetal ., 2012) .

ELIGIBILITY:
Inclusion Criteria:

1. age : from first day of life - 2 years
2. exclusively breast feeding,breast-fed infants with supplementary foods and non-breast-fed infants with supplementary foods who complain from either frequentregurgitation,vomiting,diarrhea,constipation)with/without perianal rash),bloodin stool or pallor.

Exclusion Criteria:

* Infant and child with gastrointestinal symptoms due to specific aetiology .

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of cow's milk protein allergy | baseline
  The study will assess the diagnosis of Cow's milk protein allergy (CMPA) among infant and children in Assiut University Children Hospital using skin prick test and specificserumIgE

REFERENCES:
- [Background] Celik-Bilgili S, Mehl A, Verstege A, Staden U, Nocon M, Beyer K, Niggemann B. The predictive value of specific immunoglobulin E levels in serum for the outcome of oral food challenges. Clin Exp Allergy. 2005 Mar;35(3):268-73. doi: 10.1111/j.1365-2222.2005.02150.x. PMID 15784102
- [Background] Brill H. Approach to milk protein allergy in infants. Can Fam Physician. 2008 Sep;54(9):1258-64. PMID 18791102
- [Background] Vandenplas Y, De Greef E, Devreker T. Treatment of Cow's Milk Protein Allergy. Pediatr Gastroenterol Hepatol Nutr. 2014 Mar;17(1):1-5. doi: 10.5223/pghn.2014.17.1.1. Epub 2014 Mar 31. PMID 24749081
- [Background] Sicherer SH, Noone SA, Koerner CB, Christie L, Burks AW, Sampson HA. Hypoallergenicity and efficacy of an amino acid-based formula in children with cow's milk and multiple food hypersensitivities. J Pediatr. 2001 May;138(5):688-93. doi: 10.1067/mpd.2001.113007. PMID 11343044
- [Background] Koletzko S, Niggemann B, Arato A, Dias JA, Heuschkel R, Husby S, Mearin ML, Papadopoulou A, Ruemmele FM, Staiano A, Schappi MG, Vandenplas Y; European Society of Pediatric Gastroenterology, Hepatology, and Nutrition. Diagnostic approach and management of cow's-milk protein allergy in infants and children: ESPGHAN GI Committee practical guidelines. J Pediatr Gastroenterol Nutr. 2012 Aug;55(2):221-9. doi: 10.1097/MPG.0b013e31825c9482. PMID 22569527
- [Background] Venter C, Brown T, Shah N, Walsh J, Fox AT. Diagnosis and management of non-IgE-mediated cow's milk allergy in infancy - a UK primary care practical guide. Clin Transl Allergy. 2013 Jul 8;3(1):23. doi: 10.1186/2045-7022-3-23. PMID 23835522
- [Background] NIAID-Sponsored Expert Panel; Boyce JA, Assa'ad A, Burks AW, Jones SM, Sampson HA, Wood RA, Plaut M, Cooper SF, Fenton MJ, Arshad SH, Bahna SL, Beck LA, Byrd-Bredbenner C, Camargo CA Jr, Eichenfield L, Furuta GT, Hanifin JM, Jones C, Kraft M, Levy BD, Lieberman P, Luccioli S, McCall KM, Schneider LC, Simon RA, Simons FE, Teach SJ, Yawn BP, Schwaninger JM. Guidelines for the diagnosis and management of food allergy in the United States: report of the NIAID-sponsored expert panel. J Allergy Clin Immunol. 2010 Dec;126(6 Suppl):S1-58. doi: 10.1016/j.jaci.2010.10.007. PMID 21134576